CLINICAL TRIAL: NCT06449586
Title: CMV-specific T Cell Immunity Test Indicated Prophylaxis of Letermovir After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: CMV-specific T Cell Immunity Test Indicated Prophylaxis of Letermovir After All-HSCT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Xiaoxia, Principal Investigator, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RJBMT-2024-02
Record Dates: First submitted 2024-06-01; First posted 2024-06-10 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMI-F (Experimental): Letemovir prophylaxis stops when CMV-FlowSpot >1.5.
  Interventions: Drug: Letermovir
- CMI-N (Other): Letemovir prophylaxis stopos in the first 100 days after allo-HSCT.
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — letermovir stops when CMI>1.5

SUMMARY:
To evaluate the efficacy of CMV-specific T cell immunity test in prolonged usage of letermovir for avoiding late-onset csCMVi after all-HSCT.

DETAILED DESCRIPTION:
Reactivation of cytomegalovirus (CMV) leads to significant morbidity and mortality following allogeneic hematopoietic stem cell transplantation (allo-HSCT). Letermovir (LTV) has substantially reduced the risk of clinically significant CMV infection (csCMVi) in CMV seropositive recipients of allo-HSCT. LTV discontinuation after day 100 (d100) has been reported to increase the risk of late-onset csCMVi, causing by impaired reconstitution of CMV-specific T immunity. The investigator sought to decrease the probability of CS-CMVi after letermovir withdrawal. Restoration of CMV-specific T cells is imperative for effective control of CMV reactivation following allo-HSCT. Letermovir has been found impending recovery of CMV-specific T immunity. The investigators' retrospective study has proved that lower CMV-specific CD4+ T cells (<2.01 cells/µL) at week 8 increased the risk of late-onset CMV reactivation (50.0%) compared to the higher ones (7.69%, p=0.04) in letermovir prophylaxis. Thus, the guidance of CMV-specific cell immunity is recommended in letermovir prophylaxis.

Therefore, the investigator conduct a multicenter, randomized, controlled study based on retrospective research to further explore and validate the efficacy of CMV-specific T cell immunity test guiding the prolonged usage of letermovir.

ELIGIBILITY:
Inclusion Criteria:

* first allogeneic hematopoietic stem cell transplantation;
* 18-70 years old;
* use cytomegalovirus prophylaxis with letemovir after allo-HSCT;
* CMV Ig G D+/R+;

Exclusion Criteria:

* Allergy, known hypersensitivity to letermovir tablet or injection components;
* CMV DNAemia within six months before transplantation or previous CMV disease;
* Presence of organ failure and inability to tolerate allogeneic hematopoietic stem cell transplantation;
* Second transplantation;
* Combination of immunodeficiency diseases;
* Those judged by the investigator to be unsuitable for participation in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of late-onset clinical significant CMV (cs-CMV) infection | through study completion, an average of 1 year
  Incidence of late-onset clinical significant CMV (cs-CMV) infection

SECONDARY OUTCOMES:
cumulative incidence of cs-CMV infection | through study completion, an average of 1 year
  cumulative incidence of cs-CMV infection
overall survival | through study completion, an average of 1 year
  overall survival

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Tongji Hospital of Huazhong University of Science and Technology, Wuhan, Wuhan, Hubei
  - Ruijin Hospital of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - The First Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai
  - Shanghai Liquan Hospital, Shanghai